CLINICAL TRIAL: NCT01088815
Title: A Phase II Study of Gemcitabine and Nab-Paclitaxel in Combination With GDC-0449 (Hedgehog Inhibitor) in Patients With Previously Untreated Metastatic Adenocarcinoma of the Pancreas
Brief Title: Hedgehog Inhibitors for Metastatic Adenocarcinoma of the Pancreas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Stand Up To Cancer (Other); Genentech, Inc. (Industry); Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J1013; NA_00036883 (Other: JHM IRB)
Record Dates: First submitted 2010-03-01; First posted 2010-03-17 (Estimated); Results first posted 2019-04-26 (Actual); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Metastatic Pancreatic Cancer
Keywords: Adenocarcinoma; Hedgehog; Neoplasms; Digestive System Diseases; Neoplasms by Site; Digestive System Neoplasms; Neoplasms by Histologic Type; Pancreatic Neoplasms; Pancreatic Diseases; Carcinoma
MeSH Terms: conditions — Pancreatic Neoplasms; Adenocarcinoma; Neoplasms; Digestive System Diseases; Neoplasms by Site; Digestive System Neoplasms; Neoplasms by Histologic Type; Pancreatic Diseases; Carcinoma | interventions — Gemcitabine; 130-nm albumin-bound paclitaxel; HhAntag691

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gemcitabine, nab-paclitaxel, GDC-0449 (Experimental): Gemcitabine and nab-Paclitaxel in combination with GDC-0449 (Vismodegib)
  Interventions: Drug: Gemcitabine, nab-Paclitaxel, GDC-0449

INTERVENTIONS:
Drug: Gemcitabine, nab-Paclitaxel, GDC-0449 — 1. One cycle of Gemcitabine 1000 mg/m2 and nab-Paclitaxel 125 mg/m2 on days 1, 8, and 15 (28 days cycle) then
  2. Gemcitabine 1000 mg/m2 and nab-Paclitaxel 125 mg/m2 on days 1, 8, and 15 every 28 days cycle in combination with oral GDC-0449 150 mg daily

SUMMARY:
This is an open-label, single arm, multi-center, Phase II trial to evaluate the progression free survival in patients with metastatic adenocarcinoma of the pancreas treated with a hedgehog inhibitor (GDC-0449) in combination with chemotherapy (gemcitabine and nab-Paclitaxel).

DETAILED DESCRIPTION:
The emergence of new small molecules with capacity of blocking the Hedgehog signaling pathway provides a novel therapeutic approach in pancreatic adenocarcinoma treating the primary tumor, stroma, systemic metastases and pancreatic cancer stem cells by hedgehog pathway inhibition. This phase 2 clinical trial will evaluate the progression free survival (PFS) in patients with previously untreated metastatic pancreatic adenocarcinoma. We hypothesize that the combination of cytotoxic agents (gemcitabine and nab-paclitaxel) with the Hedgehog inhibitor GDC-0449 may increase PFS.

This study includes correlative studies to attempt to understand the stem cell biology and mechanism for any observed clinical benefits with the use of Hedgehog inhibitor GDC-0449. These include changes in the hedgehog pathway and changes in pancreatic cancer stem cell markers with pre and post treatment biopsies. The safety of GDC-0449 when combined with chemotherapy gemcitabine and nab-paclitaxel will also be assessed by evaluating adverse event rate.

Following the determination of eligibility patients will receive the following treatment:

1. One cycle of Gemcitabine 1000 mg/m2 and nab-Paclitaxel 125 mg/m2 on days 1, 8, and 15 (28 days cycle) then
2. Gemcitabine 1000 mg/m2 and nab-Paclitaxel 125 mg/m2 on days 1, 8, and 15 every 28 days cycle in combination with oral GDC-0449 150 mg daily

Patients may continue on treatment regimen until they experience progressive disease or unacceptable toxicity, require palliative radiotherapy, withdraw consent or the physician feels it is not longer in their best interest to continue on treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has histologically or cytologically confirmed metastatic adenocarcinoma of the pancreas. Patients with islet cells tumors are excluded. Biopsy within 14 days of starting treatment.
2. Patient has measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >20 mm with conventional techniques or as >10 mm with spiral CT scan.
3. Patient has NOT received previous radiotherapy, surgery or chemotherapy or investigational drug therapy for the treatment of metastatic disease. If the patient received radiotherapy, chemotherapy or investigational therapy in the adjuvant setting it should be completed 3 weeks prior to enrollment. If a patient received gemcitabine in the adjuvant setting, tumor recurrence must have occurred at least six months after completing the last dose of gemcitabine
4. Age >18 years.
5. Life expectancy of greater than 1 month.
6. ECOG performance status 0 or 1 (Karnofsky >70%).
7. Patients must have adequate organ and marrow function

Exclusion Criteria:

1. Patient had received chemotherapy or radiotherapy for metastatic disease
2. Patient is receiving other investigational agents.
3. Patient has known brain metastases, unless previously treated and well controlled for at least three months (defined as clinically stable, no edema, no steroids and stable in 2 scans at least 4 weeks apart)
4. History of allergic reactions attributed to compounds of similar chemical or biologic composition to GDC-0449 or other agents used in the study.
5. Patients taking medications with narrow therapeutic indices that are metabolized by cytochrome P450 (CYP450), including warfarin sodium (Coumadin®) are ineligible.
6. Uncontrolled illness including, but not limited to, ongoing or active infection requiring IV antibiotics, symptomatic congestive heart failure not controlled with medication, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
7. Pregnant women are excluded
8. Patient has undergone a major surgery, other than diagnostic surgery (i.e. surgery done to obtain a biopsy for diagnosis without removal of an organ) within four weeks prior to Day 1 of treatment on this study.
9. History of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates use of an investigational drug or that might affect interpretation of the results of the study or render the patient at high risk from treatment complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2010-09-17 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2018-02-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Laheru, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center JHMI; Ana De Jesus-Acosta, MD, Principal Investigator — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (3):
- United States (3):
  - Translational Genomics Research Institute (TGen), Scottsdale, Arizona
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - University of Pennsylvania, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] De Jesus-Acosta A, Sugar EA, O'Dwyer PJ, Ramanathan RK, Von Hoff DD, Rasheed Z, Zheng L, Begum A, Anders R, Maitra A, McAllister F, Rajeshkumar NV, Yabuuchi S, de Wilde RF, Batukbhai B, Sahin I, Laheru DA. Phase 2 study of vismodegib, a hedgehog inhibitor, combined with gemcitabine and nab-paclitaxel in patients with untreated metastatic pancreatic adenocarcinoma. Br J Cancer. 2020 Feb;122(4):498-505. doi: 10.1038/s41416-019-0683-3. Epub 2019 Dec 20. PMID 31857726

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 98 subjects signed consents in total. 26 subjects were screen-fails
Period: Overall Study
Arm/Group | Gemcitabine, Nab-paclitaxel, GDC-0449
Started | 72
Completed | 72
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Gemcitabine, Nab-paclitaxel, GDC-0449
Number analyzed (Participants) | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 40
  >=65 years | 32
Age, Continuous [Mean (Full Range); unit: years] | 62.05 [18 to 100]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 71
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 64
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 72

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival With the Combination of GDC-0449 With Gemcitabine and Nab-paclitaxel.
Description: Number of months from time first therapy received to the earliest documented disease progression or death from any cause.
Time Frame: 6 years
Population: Data for this outcome measure was evaluable in only in 67/72 participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Gemcitabine, Nab-paclitaxel, GDC-0449
Number analyzed (Participants) | 67
months | 5.42 [4.37 to 6.97]

2. Primary Outcome: Safety of Combination Therapy in Patients With Metastatic Adenocarcinoma of the Pancreas as Assessed by Number of Grade 3 or 4 Adverse Events
Description: Number of grade 3 or 4 adverse events as defined by National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI CTCAE v4.0) that occur after Cycle 2, Day 1
Time Frame: 6 years
Measure: Number; unit: Grade 3/4 adverse events
Arm/Group | Gemcitabine, Nab-paclitaxel, GDC-0449
Number analyzed (Participants) | 72
Grade 3/4 adverse events | 104

3. Secondary Outcome: Efficacy of Combination of GDC-0449 With Gemcitabine and Nab-Paclitaxel as Assessed by Overall Survival
Description: Total number of months alive.
Time Frame: 6 years
Population: Data was evaluable in only 67/72 participants for this outcome measure
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Gemcitabine, Nab-paclitaxel, GDC-0449
Number analyzed (Participants) | 67
months | 9.79 [7.85 to 10.97]

4. Secondary Outcome: Efficacy of Combination of GDC-0449 With Gemcitabine and Nab-Paclitaxel as Assessed by Tumor Response
Description: Number of participants with complete (CR) or partial (PR) response as defined by RECIST criteria.
Time Frame: 6 years
Population: Data was evaluable in only 67/72 participants for this outcome measure
Measure: Count of Participants; unit: Participants
Arm/Group | Gemcitabine, Nab-paclitaxel, GDC-0449
Number analyzed (Participants) | 67
Participants
  CR | 1
  PR | 26

5. Secondary Outcome: Efficacy of Combination of GDC-0449 With Gemcitabine and Nab-Paclitaxel as Assessed by Changes in Pancreatic Cancer Stem Cell
Description: Change in number of Pancreatic cancer stem cells in tissue and peripheral blood in tissue biopsy and peripheral blood.
Time Frame: 6 years
Population: Peripheral blood data was collected from only 57/72 participants. Tissue biopsy data was not evaluable for analysis due to inadequate biopsy samples for all 23/72 participants who underwent biopsy
Measure: Mean (Standard Deviation); unit: cells
Arm/Group | Gemcitabine, Nab-paclitaxel, GDC-0449
Number analyzed (Participants) | 72
cells
  peripheral blood: number analyzed (Participants) | 57
  peripheral blood | 27.0 (4.0)
  tissue biopsy: number analyzed (Participants) | 0

6. Secondary Outcome: Efficacy of Combination of GDC-0449 With Gemcitabine and Nab-Paclitaxel as Assessed by Hedgehog Signaling Pathway Downregulation
Description: Hedgehog signaling pathway downregulation as measured by Gli-1 and Patch expression
Time Frame: 6 years
Population: Data was not collected for this outcome measure.
Arm/Group | Gemcitabine, Nab-paclitaxel, GDC-0449
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 6 years
Arm/Group | Gemcitabine, Nab-paclitaxel, GDC-0449
All-Cause Mortality (participants affected / at risk) | 64/72
Serious Adverse Events (participants affected / at risk) | 46/72
Other Adverse Events (participants affected / at risk) | 72/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine, Nab-paclitaxel, GDC-0449 (N=72)
Abdominal Distension (Blood and lymphatic system disorders) | 1 (1)
Febrile Neutropenia (Blood and lymphatic system disorders) | 2 (2)
Abdominal Pain (Gastrointestinal disorders) | 2 (2)
Acute Kidney Injury (Renal and urinary disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 3 (3)
Ascites (Gastrointestinal disorders) | 1 (1)
Atrial Fibrillation (Cardiac disorders) | 1 (1)
Blood Bilirubin Increased (Blood and lymphatic system disorders) | 1 (1)
Blood/Lymph Disorder (Blood and lymphatic system disorders) | 1 (1)
Death (General disorders) | 5 (5)
Dehyrdation (Metabolism and nutrition disorders) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Duodenal Obstruction (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Fever (General disorders) | 8 (9)
Gallbladder Infection (Gastrointestinal disorders) | 1 (1)
Gastroparesis (Gastrointestinal disorders) | 1 (1)
General Disorders/Administration Site (General disorders) | 1 (1)
GI disorders (Gastrointestinal disorders) | 2 (3)
Heart Failure (Cardiac disorders) | 1 (1)
Hematoma (Vascular disorders) | 2 (2)
Hepatobil Disorders (Hepatobiliary disorders) | 4 (4)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2)
Hypotension (Vascular disorders) | 2 (2)
Ileus (Eye disorders) | 1 (2)
Infestion/Infestation-Other (Infections and infestations) | 2 (2)
Investigations-Other (Investigations) | 4 (4)
Kidney Infection (Renal and urinary disorders) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Neutrophil Count Decreased (Investigations) | 2 (2)
Obstruction Gastric (Gastrointestinal disorders) | 1 (1)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Pericardial Effusion (Cardiac disorders) | 1 (1)
Platelet Count Decreased (Investigations) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Respiratory/Thoracic/Mediastinal Disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sepsis (Infections and infestations) | 6 (6)
Skin Infection (Skin and subcutaneous tissue disorders) | 4 (4)
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 (1)
Splenic Infection (Infections and infestations) | 1 (1)
Stroke (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (2)
Thromboembolic (Vascular disorders) | 4 (4)
Upper GI Hemorrhage (Gastrointestinal disorders) | 2 (4)
Urinary Tract Obstruction (Renal and urinary disorders) | 1 (1)
Vascular Access Complication (Vascular disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Wound Infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gemcitabine, Nab-paclitaxel, GDC-0449 (N=72)
Abdominal Distension (Gastrointestinal disorders) | 5 (5)
Abdominal Pain (Gastrointestinal disorders) | 19 (23)
Agitation (Psychiatric disorders) | 1 (1)
Alkaline Phosphatase Increased (Investigations) | 23 (38)
Alkalosis (Metabolism and nutrition disorders) | 1 (1)
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 46 (58)
ALT Increased (Investigations) | 34 (60)
Anal Hemorrhage (Gastrointestinal disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 56 (232)
Anorexia (Metabolism and nutrition disorders) | 26 (37)
Anxiety (Psychiatric disorders) | 7 (7)
APTT Prolonged (Investigations) | 4 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Ascites (Gastrointestinal disorders) | 12 (14)
AST Increased (Investigations) | 35 (53)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 9 (9)
Atrial Fibrillation (Cardiac disorders) | 1 (1)
Atrial Flutter (Cardiac disorders) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 6 (6)
Bile Duct Stenosis (Hepatobiliary disorders) | 1 (1)
Bloating (Gastrointestinal disorders) | 3 (3)
Blood Bilirubin Increased (Blood and lymphatic system disorders) | 12 (19)
Blood/Lymph Disorder (Blood and lymphatic system disorders) | 4 (4)
Breast Pain (Reproductive system and breast disorders) | 1 (1)
Bruising (Skin and subcutaneous tissue disorders) | 5 (5)
Bullous Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Cardiac Troponin I Increased (Cardiac disorders) | 1 (1)
Cardiac Troponin T Increased (Cardiac disorders) | 1 (1)
CD34 Lymphocytes Decreased (Investigations) | 1 (1)
Chest Pain - Cardiac (Cardiac disorders) | 1 (1)
Chest Wall Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Chills (General disorders) | 14 (15)
Concentration Impairment (Psychiatric disorders) | 1 (1)
Confusion (Psychiatric disorders) | 4 (7)
Constipation (Gastrointestinal disorders) | 17 (21)
Cough (Respiratory, thoracic and mediastinal disorders) | 17 (19)
CPK Increased (Investigations) | 1 (1)
Creatinine Increased (Investigations) | 9 (11)
Dehydration (Metabolism and nutrition disorders) | 11 (37)
Depression (Psychiatric disorders) | 6 (6)
Diarrhea (Gastrointestinal disorders) | 30 (43)
Dizziness (Nervous system disorders) | 18 (18)
Dry Eye (Eye disorders) | 1 (1)
Dry Mouth (Gastrointestinal disorders) | 6 (8)
Dry Skin (Skin and subcutaneous tissue disorders) | 4 (5)
Duodenal Perforation (Gastrointestinal disorders) | 1 (1)
Dysarthria (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 53 (74)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
dysphagia (Gastrointestinal disorders) | 2 (3)
Dysphasia (Nervous system disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 23 (30)
ECG QT Corrected int prolong (Cardiac disorders) | 1 (1)
Edema Face (General disorders) | 1 (1)
Edema Limbs (General disorders) | 28 (52)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 10 (10)
Erythema Multiforme (Skin and subcutaneous tissue disorders) | 3 (5)
Erythroderma (Skin and subcutaneous tissue disorders) | 1 (3)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Extrapyramidal Disorder (Nervous system disorders) | 1 (1)
Eye Disorder - Other (Eye disorders) | 2 (2)
Facial Nerve Disorder (Nervous system disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Fatigue (General disorders) | 49 (97)
Febrile Neutropenia (Blood and lymphatic system disorders) | 2 (2)
Fecal incontinence (Gastrointestinal disorders) | 1 (1)
Fever (General disorders) | 22 (38)
Flank Pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Flatulence (Gastrointestinal disorders) | 6 (6)
Flu like symptoms (General disorders) | 12 (16)
Fracture (Musculoskeletal and connective tissue disorders) | 2 (2)
Gait Disturbance (General disorders) | 4 (5)
Gastric Ulcer (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 2 (2)
General disorders/admin site conditions (General disorders) | 5 (5)
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 6 (8)
Genital Edema (Reproductive system and breast disorders) | 3 (3)
GERD (Gastrointestinal disorders) | 3 (3)
GI disorders - other (Gastrointestinal disorders) | 11 (14)
Hallucinations (Psychiatric disorders) | 1 (1)
Headache (Nervous system disorders) | 6 (8)
Hematoma (Vascular disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 2 (2)
Hemoglobinuria (Renal and urinary disorders) | 1 (1)
Hemorrhoidal Hemorrhage (Gastrointestinal disorders) | 2 (2)
Hemorrhoids (Gastrointestinal disorders) | 1 (1)
Hepatobil disorders - other (Hepatobiliary disorders) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 31 (65)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 12 (15)
Hypermagnesemia (Metabolism and nutrition disorders) | 5 (6)
Hypertension (Vascular disorders) | 2 (3)
Hypoalbuminemia (Metabolism and nutrition disorders) | 33 (91)
Hypocalcemia (Metabolism and nutrition disorders) | 29 (60)
Hypoglycemia (Metabolism and nutrition disorders) | 3 (5)
Hypokalemia (Metabolism and nutrition disorders) | 20 (37)
Hypomagnesemia (Metabolism and nutrition disorders) | 9 (15)
Hyponatremia (Metabolism and nutrition disorders) | 24 (47)
Hypophosphatemia (Metabolism and nutrition disorders) | 11 (19)
Hypotension (Vascular disorders) | 12 (19)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Infections/Infestactions - Other (Infections and infestations) | 10 (13)
Infusion site extravasation (Injury, poisoning and procedural complications) | 1 (1)
Injection site reaction (Injury, poisoning and procedural complications) | 1 (1)
INR Increased (Investigations) | 8 (10)
Insomnia (Psychiatric disorders) | 6 (6)
Intracranial hemorrhage (Nervous system disorders) | 1 (1)
Investigations-Other, specify (Investigations) | 8 (12)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Lethargy (Nervous system disorders) | 2 (2)
Leukocytosis (Blood and lymphatic system disorders) | 3 (3)
Lipase increased (Investigations) | 2 (3)
Localized edema (General disorders) | 5 (5)
Lung infection (Infections and infestations) | 4 (4)
Lymphocyte count decreased (Investigations) | 41 (175)
Lymphocyte count increased (Investigations) | 4 (4)
Malaise (General disorders) | 2 (4)
Metabolism/nutrition disorders-Other (Metabolism and nutrition disorders) | 1 (1)
Musculoskeletal and connective tissue disorder (Musculoskeletal and connective tissue disorders) | 12 (24)
Mucosal infection (Infections and infestations) | 3 (4)
Mucositis oral (Gastrointestinal disorders) | 8 (9)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 9 (12)
Nail discoloration (Skin and subcutaneous tissue disorders) | 4 (4)
Nail Loss (Skin and subcutaneous tissue disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 41 (56)
Neck Edema (Skin and subcutaneous tissue disorders) | 1 (1)
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Nervous system disorders - other (Nervous system disorders) | 6 (8)
Neutrophil count decreased (Investigations) | 41 (138)
Non-Cardiac Chest Pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Oculomotor nerve disorder (Nervous system disorders) | 1 (1)
Oral dysesthesia (Gastrointestinal disorders) | 1 (1)
Oral Pain (Gastrointestinal disorders) | 1 (1)
Pain (General disorders) | 11 (12)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (7)
Paresthesia (Nervous system disorders) | 9 (17)
Pericardial effusion (Cardiac disorders) | 6 (7)
Periodontal disease (Gastrointestinal disorders) | 1 (2)
Periorbital edema (Skin and subcutaneous tissue disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 16 (27)
Peripheral sensory neuropathy (Nervous system disorders) | 36 (77)
Photophobia (Eye disorders) | 1 (1)
Platelet count decreased (Investigations) | 44 (155)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 14 (15)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 10 (10)
Presyncope (Nervous system disorders) | 1 (2)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Prostatic obstruction (Reproductive system and breast disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 5 (6)
Pruritus (Skin and subcutaneous tissue disorders) | 12 (14)
Psych disorders-Other, spec (Psychiatric disorders) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 30 (36)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 11 (19)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (3)
Renal/urinary disorders-Other (Renal and urinary disorders) | 4 (5)
Repro system/breast ds-Oth (Reproductive system and breast disorders) | 1 (1)
Resp/thoracic/mediastinal ds (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Restlessness (Nervous system disorders) | 1 (1)
Right ventricular dysfunction (Cardiac disorders) | 1 (2)
Scalp pain (Skin and subcutaneous tissue disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Sinusitis (Infections and infestations) | 5 (5)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 3 (3)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Skin infection (Infections and infestations) | 7 (11)
Skin ulceration (Skin and subcutaneous tissue disorders) | 2 (2)
Skin/subq tissue ds-Other (Skin and subcutaneous tissue disorders) | 9 (17)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (2)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Stomach Pain (Gastrointestinal disorders) | 2 (3)
Syncope (Cardiac disorders) | 2 (2)
Thromboembolic event (Vascular disorders) | 16 (17)
Tremor (Nervous system disorders) | 1 (1)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 3 (5)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 2 (2)
Urinary tract infection (Renal and urinary disorders) | 4 (4)
Urine discoloration (Renal and urinary disorders) | 1 (1)
Uterine hemorrhage (Reproductive system and breast disorders) | 1 (1)
Vasc disorders-Other, spec (Vascular disorders) | 3 (3)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 30 (40)
Watering eyes (Eye disorders) | 1 (1)
Weight gain (Investigations) | 3 (3)
Weight loss (Investigations) | 16 (26)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (2)
White blood cell decreased (Investigations) | 51 (285)
Wound infection (Infections and infestations) | 2 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-12-04): https://cdn.clinicaltrials.gov/large-docs/15/NCT01088815/Prot_SAP_000.pdf